CLINICAL TRIAL: NCT04395872
Title: Psychiatric Consultation for COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Jonghun Lee, M.D., Ph. D., Daegu Catholic University Medical Center
Other Study IDs: CR-20-062
Record Dates: First submitted 2020-05-08; First posted 2020-05-20 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Covid19; Psychiatric Problem; Isolation, Social
Keywords: COVID-19; consultation
MeSH Terms: conditions — COVID-19; Social Isolation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Among patients who were confirmed as COVID-19 and admitted to the COVID-19 management ward of Daegu Catholic University Hospital, patients who were consulted by the Department of psychiatry was selected as participants. Socio-demographic information, medical severity (oxygen saturation, chest x-ray readings, medication being administered), clinical psychological scale (PHQ-9, GAD-7, PC-PTSD-5, AIS, P4, SF-36, SCL-90-R). were collected from participants. It evaluates whether there is a difference in the psychological scale according to the difference in participants' sociodemographic status and medical severity, and evaluates the effectiveness of psychiatric counseling by comparing clinical psychological measures before and after referral to department of psychiatry.
  Interventions: Behavioral: Psychiatric counseling

INTERVENTIONS:
Behavioral: Psychiatric counseling — Patients who are admitted to the COVID-19 care unit of the Catholic University of Daegu Hospital are subject to consultation with the psychiatrist. By retrospectively reviewing the medical records of the request and the results of the subjects, We collected Socio-demographic information, medical severity (oxygen saturation, chest x-ray readings, medication being administered), clinical psychological scale (PHQ-9, GAD-7, PC-PTSD-5, AIS, P4, SF-36, SCL-90-R) This study evaluates whether there is a difference in psychological scale according to differences in socio-demographic status and medical severity, and compares psychological psychological measures before and after referral to mental health medicine to evaluate the effectiveness of psychiatric counseling.

SUMMARY:
In this study, the content and results of the psychiatric consultation on patients in Corona Care Ward were verified retroactively, and the effects of COVID-19 patients' emotional state and psychological support and crisis intervention were assessed on their emotional state.

Patients who are admitted to the COVID-19 care unit of the Catholic University of Daegu Hospital are subject to consultation with the psychiatrist. By retrospectively reviewing the medical records of the request and the results of the subjects, We collected Socio-demographic information, medical severity (oxygen saturation, chest x-ray readings, medication being administered), clinical psychological scale (PHQ-9, GAD-7, PC-PTSD-5, AIS, P4, SF-36, SCL-90-R) This study evaluates whether there is a difference in psychological scale according to differences in socio-demographic status and medical severity, and compares psychological measures before and after referral to mental health medicine to evaluate the effectiveness of psychiatric counseling.

DETAILED DESCRIPTION:
Patients and medical workers in the event of an pandemic infectious disease usually experience extreme fear, which requires quick and immediate management of mental health. In 2015, the risk of post-traumatic stress disorder in isolated MERS patients and medical staff was very high. Even 4 ~ 6 months after the quarantine was over, anxiety was still lingering in 3% percent of patients and anger in 6.4 % of patients. The negative emotions and stress experienced by the medical staff for MERS patients were characterized by such events as mistakes and delays caused by communication problems. Also, people who were not infected with MERS experienced anxiety at 7.6 percent and anger at 16.6 percent during the quarantine period.Therefore, the need for psychological support for infected patients, isolated people, medical staff and the general public had been proposed during these infectious disease fad periods since MERS. Since the recent spread of coronavirus infection-19 (COVID-19) that began in Wuhan, China in December 2019, thousands of confirmed and dozens of deaths have been reported in South Korea and the number is on the rise. Thus, quarantine measures are currently being taken in Korea to reduce and treat the spread of COVID-19. Thus, psychological support and crisis intervention are needed in the early stages of stressful times to reduce anxiety, depression and post-traumatic stress disorder. In response, Daegu Catholic university hospital psychiatry department conducted active psychiatric counseling for medical patients who are hospitalized in Corona's management hospital for confirmation of coronavirus infection. In this study, the content and results of the psychiatric consultation on patients in Corona Care Ward were verified retroactively, and the effects of COVID-19 patients' emotional state and psychological support and crisis intervention were assessed on their emotional state.

Patients who are admitted to the COVID-19 care unit of the Catholic University of Daegu Hospital are subject to consultation with the psychiatrist. By retrospectively reviewing the medical records of the request and the results of the subjects, We collected Socio-demographic information, medical severity (oxygen saturation, chest x-ray readings, medication being administered), clinical psychological scale (PHQ-9, GAD-7, PC-PTSD-5, AIS, P4, SF-36, SCL-90-R) This study evaluates whether there is a difference in psychological scale according to differences in socio-demographic status and medical severity, and compares psychological psychological measures before and after referral to mental health medicine to evaluate the effectiveness of psychiatric counseling.

ELIGIBILITY:
Inclusion Criteria:

1. Patient admitted to the COVID-19 management ward of Daegu Catholic University Hospital
2. Patients who were consulted with a psychiatrist by a physician.

Exclusion Criteria:

1. When the subject is accompanied by a serious physical or neurological condition
2. In case of brain damage or concussion with loss of consciousness at the time of treatment
3. When it is difficult to understand psychological intervention due to the apparent decrease in intelligence at the time of treatment
4. When it is difficult to understand psychological intervention and follow examination instructions due to noticeable sensory damage such as hearing and vision at the time of treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been confirmed as COVID-19 and admitted to the management ward, and consulted with a psychiatrist by a physician.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2020-05-28 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of PHQ-9 (Patient Health Questionnaire-9) | On admission and at the time of discharge, on average 2 months
  for assess depressive symptom
Change of GAD-7 (Patient Health Questionnaire-9) | On admission and at the time of discharge, on average 2 months
  for assess anxiety symptom
Change of PC-PTSD-5 (Primary Care PTSD Screen for DSM-5) | On admission and at the time of discharge, on average 2 months
  for assess PTSD symptom
Change of AIS (Athens Insomnia Scale) | On admission and at the time of discharge, on average 2 months
  for assess insomnia
Change of P4 (P4 Suicidality Screener) | On admission and at the time of discharge, on average 2 months
  for assess suicidal idea
Change of SF-36 (Short Form Health Survey Questionnaire) | On admission and at the time of discharge, on average 2 months
  for assess health associated QoL

SECONDARY OUTCOMES:
Change of SCL-90-R | On admission and at the time of discharge, on average 2 months
  for assess other psychiatric symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jonghun Lee, M.D., ph.D., Principal Investigator — Daegu Catholic University Medical Center

IPD SHARING:
Plan to Share IPD: No
Data will be shared on request for proper reason.

REFERENCES:
- [Background] Folkman S, Greer S. Promoting psychological well-being in the face of serious illness: when theory, research and practice inform each other. Psychooncology. 2000 Jan-Feb;9(1):11-9. doi: 10.1002/(sici)1099-1611(200001/02)9:13.0.co;2-z. PMID 10668055
- [Background] Kang L, Li Y, Hu S, Chen M, Yang C, Yang BX, Wang Y, Hu J, Lai J, Ma X, Chen J, Guan L, Wang G, Ma H, Liu Z. The mental health of medical workers in Wuhan, China dealing with the 2019 novel coronavirus. Lancet Psychiatry. 2020 Mar;7(3):e14. doi: 10.1016/S2215-0366(20)30047-X. Epub 2020 Feb 5. No abstract available. PMID 32035030
- [Background] Lee SM, Kang WS, Cho AR, Kim T, Park JK. Psychological impact of the 2015 MERS outbreak on hospital workers and quarantined hemodialysis patients. Compr Psychiatry. 2018 Nov;87:123-127. doi: 10.1016/j.comppsych.2018.10.003. Epub 2018 Oct 13. PMID 30343247
- [Background] Maunder R, Hunter J, Vincent L, Bennett J, Peladeau N, Leszcz M, Sadavoy J, Verhaeghe LM, Steinberg R, Mazzulli T. The immediate psychological and occupational impact of the 2003 SARS outbreak in a teaching hospital. CMAJ. 2003 May 13;168(10):1245-51. PMID 12743065
- [Background] Okusaga O, Yolken RH, Langenberg P, Lapidus M, Arling TA, Dickerson FB, Scrandis DA, Severance E, Cabassa JA, Balis T, Postolache TT. Association of seropositivity for influenza and coronaviruses with history of mood disorders and suicide attempts. J Affect Disord. 2011 Apr;130(1-2):220-5. doi: 10.1016/j.jad.2010.09.029. Epub 2010 Oct 27. PMID 21030090
- [Background] Park SC, Park YC. Mental Health Care Measures in Response to the 2019 Novel Coronavirus Outbreak in Korea. Psychiatry Investig. 2020 Feb;17(2):85-86. doi: 10.30773/pi.2020.0058. Epub 2020 Feb 25. No abstract available. PMID 32093458
- [Background] Xiang YT, Yang Y, Li W, Zhang L, Zhang Q, Cheung T, Ng CH. Timely mental health care for the 2019 novel coronavirus outbreak is urgently needed. Lancet Psychiatry. 2020 Mar;7(3):228-229. doi: 10.1016/S2215-0366(20)30046-8. Epub 2020 Feb 4. No abstract available. PMID 32032543
- [Background] Xiao C. A Novel Approach of Consultation on 2019 Novel Coronavirus (COVID-19)-Related Psychological and Mental Problems: Structured Letter Therapy. Psychiatry Investig. 2020 Feb;17(2):175-176. doi: 10.30773/pi.2020.0047. Epub 2020 Feb 25. No abstract available. PMID 32093461
- [Background] Zhou X. Psychological crisis interventions in Sichuan Province during the 2019 novel coronavirus outbreak. Psychiatry Res. 2020 Apr;286:112895. doi: 10.1016/j.psychres.2020.112895. Epub 2020 Feb 26. No abstract available. PMID 32120170